CLINICAL TRIAL: NCT01469533
Title: Changes in Pressure Pain Thresholds and Basal Electromyographic Activities Following Spinal Mechanical Manipulation in Asymptomatic Subjects
Brief Title: Pressure Pain Thresholds and Basal Electromyographic Activities Following Spinal Mechanical Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RenJiH-2011020
Record Dates: First submitted 2011-11-03; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Pain
Keywords: Spine; Manipulation; Pain Threshold; Electromyography.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): The experimental group receives the real spinal mechanical manipulation.
  Interventions: Other: Spinal mechanical manipulation intervention
- control group (Sham Comparator): The control group receives the sham-manipulation procedure.
  Interventions: Other: Sham manipulation intervention

INTERVENTIONS:
Other: Spinal mechanical manipulation intervention — Subjects in experimental group are assessed through use of the Activator Methods (AM) assessment protocol. Spinal adjustment of the indicated pelvis, sacrum and lumbar spine is performed through the use of spinal mechanical manipulation. In this study leg length analysis only uses Position #1 and Position #2. Mechanical manipulation is delivered with the Activator Ⅳ Adjusting Instrument (AAI Ⅳ; Activator Methods International, Ltd, Phoenix, AZ) set in the maximal force setting 4, as it is used in routine clinical practice. The Activator Ⅳ delivers a very short duration (<5 ms) force-time impulse with a peak force magnitude of approximately 176N.
  Other Names: Activator methods maximal setting
  Arms: experimental group
Other: Sham manipulation intervention — Subjects in the control group receive a protocol identical to that described above, with the following exception: a sham mechanical thrust is delivered during the AM protocol. The sham procedure is accomplished by setting the expansion control knob on the Activator Ⅱ to the zero (off) position. The expansion control is used to adjust the spring compression and thus the amount of excursion of the instruments' stylus. In the zero position, no excursion of the stylus occurs, although the same clicking sound that the instrument produces during normal use is heard after manual activation of the mechanical trigger.
  Other Names: Activator methods zero setting
  Arms: control group

SUMMARY:
The purpose of this study is to investigate if the application of spinal mechanical manipulation on low back region resulted in changes in pressure pain thresholds (PPT) in asymptomatic subjects and the extent of the hypoalgesia; whether it is local, regional or systemic. Simultaneously, the investigators are to further explore the phenomenon of reduced sEMG activity after spinal mechanical manipulation to better understand the immediate effects of mechanical manipulation on low back region.

DETAILED DESCRIPTION:
Spinal manipulation (SM) is used by clinicians for the treatment of several chronic pain conditions. The effectiveness of different spinal manipulations targeted at the lumbar spine in patients with low back pain is supported by an increasing number of high-quality randomized clinical trials1and systematic reviews. Although these techniques have shown some effectiveness in clinical practice, most of clinical studies solely investigated the effects of spinal manipulation on overall reports of pain and function and the underlying mechanisms by which manipulation produce clinical effects remain largely unknown.

The neurophysiologic mechanisms by which manipulation inhibits pain, however, are matters of speculation and still under investigation. Proposed hypotheses have suggested that manipulation has the potential to remove the source of mechanical pain or induce stimulus-produced analgesia. Spinal manipulation induces sufficient force to simultaneously activate both superficial and deep somatic mechanoreceptors, proprioceptors, and nociceptors. The effect of this stimulation is a strong afferent segmental barrage of spinal cord sensory neurons, capable of altering the pattern of afferent input to the central nervous system and inhibiting the central transmission of pain. Other suggested mechanisms have been the activation of the endogenous opiate system, the alteration of the chemical mediators or the effects of joint cavitation. An understanding of the mechanism by which manipulations cause a hypoalgesic response is subject to further research and is currently far from complete. A review of the literature found several studies exploring immediate changes in mechanical pain sensitivity provoked by spinal manipulative procedures. Mobilisation/manipulation to the cervical spine has been shown to provide a hypoalgesic effect as measured by pressure pain thresholds (PPTs) in patients suffering from mechanical neck pain and lateral epicondylalgia. A hypoalgesic effect has also been demonstrated following mobilization to peripheral joints in the upper and lower limbs. Mobilizations to the lumbar spine have been shown to produce an immediate and significant widespread hypoalgesic effect in asymptomatic subjects However, Perry et al. that found unilateral mobilizations on the lumbar spine respectively had side specific response.

Besides analgesic effect, it has been presented spinal manipulation can reduce the increased resting muscle tone or spasm, which can be monitored by surface electromyography (sEMG). If the presence of a hypertonic muscle is functionally associated with a spinal dysfunction that is correctable by SM, it would consequently follow that the associated higher EMG level would diminish after appropriate SM. In a descriptive study DeVocht JW et al. found that manipulation induces an immediate change, usually a reduction, in resting EMG level in patients with low back pain. Herzog J reported the observation of a single but very dramatic decrease in resting EMG activity in thoracic musculature within 1 second of SM. One possible segmental mechanism could be that the manipulation may induce a reflex muscle relaxation by modifying proprioceptive group 1 and 2 afferents. However, few randomly controlled trials have directly investigated the effect of spinal mechanical manipulation on basal electromyographic activity (BEA) in asymptomatic subjects.

Spinal mechanical manipulation has been widely used in clinical manual therapy. However, because mechanical thrusts usually produce no cavitations, whether mechanical techniques produce the same hypoalgesic effects and muscle relaxation as manual techniques remains untested. To further elucidate the physiologic mechanisms associated with spinal mechanical manipulation, it is essential to investigate its effects in asymptomatic individuals who do not have any active central sensitization. In fact, recent studies have supported the use of asymptomatic subjects in studies related to neurophysiological mechanisms of spinal manipulations. Further research is therefore required to clarify if there is a hypoalgesic effect or muscle relaxation in response to spinal mechanical manipulation in the lumbar region in asymptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic volunteers
* age from 18 to 60 years

Exclusion Criteria:

* aversion to manual contact
* symptoms in the low back or lower extremities
* previous history of spine surgery
* receiving any manual therapy within the past 1 month before the study
* any contraindication to manipulation
* regular use of analgesic or anti-inflammatory drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold assessment | within 10 minutes immediately after manipulation
  A mechanical pressure algometer (Wagner, Greenwich, CT) is used to measure PPT levels. Participants report to stop the pressure stimulation immediately when the sensation turnes from pressure to pain. The L5-S1 zygapophyseal is chosen as a landmark local to the manipulation. The L5 dermatome is chosen to measure the extent of any hypoalgesic response. The first dorsal interossei in the hand is selected to evaluate if there was a systemic response to the manipulation.

SECONDARY OUTCOMES:
Basal electromyographic activity | within 10 minutes immediately after manipulation
  Basal electromyographic activity (BEA) of paraspinal muscles is measured using a BioGraph@ surface electromyography with Infiniti software Systems version 1.51B (Thought Technology, Montreal, Quebec). Electrodes are 2.25-in (5.72cm) triodes, disposable, and adhesive with Ag/AgCl snaps. The electrodes are placed 30mm from the spinous process of the fourth lumbar vertebra (L4) and 10mm from the spinous process of the fifth cervical vertebra (C5). The signal is selected for 10 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangrui Wang, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Giles LG, Muller R. Chronic spinal pain: a randomized clinical trial comparing medication, acupuncture, and spinal manipulation. Spine (Phila Pa 1976). 2003 Jul 15;28(14):1490-502; discussion 1502-3. doi: 10.1097/00007632-200307150-00003. PMID 12865832
- [Background] Lawrence DJ, Meeker W, Branson R, Bronfort G, Cates JR, Haas M, Haneline M, Micozzi M, Updyke W, Mootz R, Triano JJ, Hawk C. Chiropractic management of low back pain and low back-related leg complaints: a literature synthesis. J Manipulative Physiol Ther. 2008 Nov-Dec;31(9):659-74. doi: 10.1016/j.jmpt.2008.10.007. PMID 19028250
- [Background] Boal RW, Gillette RG. Central neuronal plasticity, low back pain and spinal manipulative therapy. J Manipulative Physiol Ther. 2004 Jun;27(5):314-26. doi: 10.1016/j.jmpt.2004.04.005. PMID 15195039
- [Background] Cramer G, Budgell B, Henderson C, Khalsa P, Pickar J. Basic science research related to chiropractic spinal adjusting: the state of the art and recommendations revisited. J Manipulative Physiol Ther. 2006 Nov-Dec;29(9):726-61. doi: 10.1016/j.jmpt.2006.09.003. PMID 17142166
- [Background] Vernon H. Qualitative review of studies of manipulation-induced hypoalgesia. J Manipulative Physiol Ther. 2000 Feb;23(2):134-8. doi: 10.1016/s0161-4754(00)90084-8. PMID 10714544
- [Background] de Camargo VM, Alburquerque-Sendin F, Berzin F, Stefanelli VC, de Souza DP, Fernandez-de-las-Penas C. Immediate effects on electromyographic activity and pressure pain thresholds after a cervical manipulation in mechanical neck pain: a randomized controlled trial. J Manipulative Physiol Ther. 2011 May;34(4):211-20. doi: 10.1016/j.jmpt.2011.02.002. Epub 2011 Mar 21. PMID 21621722
- [Background] Fernandez-Carnero J, Fernandez-de-las-Penas C, Cleland JA. Immediate hypoalgesic and motor effects after a single cervical spine manipulation in subjects with lateral epicondylalgia. J Manipulative Physiol Ther. 2008 Nov-Dec;31(9):675-81. doi: 10.1016/j.jmpt.2008.10.005. PMID 19028251
- [Background] DeVocht JW, Pickar JG, Wilder DG. Spinal manipulation alters electromyographic activity of paraspinal muscles: a descriptive study. J Manipulative Physiol Ther. 2005 Sep;28(7):465-71. doi: 10.1016/j.jmpt.2005.07.002. PMID 16182019
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Cleland JA, Rodriguez-Blanco C, Alburquerque-Sendin F. Changes in pressure pain thresholds over C5-C6 zygapophyseal joint after a cervicothoracic junction manipulation in healthy subjects. J Manipulative Physiol Ther. 2008 Jun;31(5):332-7. doi: 10.1016/j.jmpt.2008.04.006. PMID 18558274